CLINICAL TRIAL: NCT03439709
Title: Multicenter Evaluation of the Effect of Upfront Radiosurgery on Residual Growth Hormone-secreting Pituitary Adenoma From an Endocrinological Point of View (MERGE Study): a Randomized, Phase 3 Trial
Brief Title: Multicenter Evaluation of the Effect of Upfront Radiosurgery on Residual Growth Hormone-secreting Pituitary Adenoma
Acronym: MERGE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2017-11-091-002
Record Dates: First submitted 2018-02-01; First posted 2018-02-20 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Acromegaly Due to Pituitary Adenoma
Keywords: acromegaly; pituitary adenoma; gamma knife radiosurgery; adjuvant treatment
MeSH Terms: conditions — Growth Hormone-Secreting Pituitary Adenoma; Acromegaly; Pituitary Neoplasms | interventions — Radiosurgery; lanreotide; Solutions; Injections

STUDY DESIGN:
Intervention Model Description: The patients with acromegaly due to growth hormone secreting pituitary adenoma who receive primary surgical resection and fail to achieve endocrinologic remission at 3 months after surgical resection are enrolled. They are devided into two groups; One consists of patients underwent upfront stereotactic radiosurgery combinated with standard drug therapy, and another group consists of patients receiving only standard drug therapy.
Masking Description: Technically, the procedure of gamma knife radiosurgery includes fixating stereotactic frame on the head of patients. Therefore, It is not possible to keep masking for participants and other investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Gamma knife radiosurgery (Leksell Gamma Knife, Elekta AB, Stockholm, Sweden) is used for intervention. Administration of standard medical therapy using Lanreotide 60 mg concurrently starts with radiosurgery
  Interventions: Radiation: Gamma knife radiosurgery; Drug: Lanreotide 60Mg Solution for Injection
- control (Active Comparator): Without radiosurgery, standard medical therapy (Lanreotide 60Mg Solution for Injection) same with interventional group is applied
  Interventions: Drug: Lanreotide 60Mg Solution for Injection

INTERVENTIONS:
Radiation: Gamma knife radiosurgery — Minimum 25 Gy of marginal dose is applied for residual tumor or resection cavity. Depending on the size of tumor, the dose can be varied.
  Arms: intervention
Drug: Lanreotide 60Mg Solution for Injection — Lanreotide injection.

SUMMARY:
In this study, the investigators hypothesize that upfront gamma knife radiosurgery with drug therapy is superior in the treatment of growth hormone-secreting pituitary tumors after primary surgical treatment compared with the drug therapy alone. This study can provide useful clinical information in the treatment of patients with acromegaly.

DETAILED DESCRIPTION:
Acromegaly is often caused by growth hormone (GH)-secreting pituitary adenoma and causes anatomic changes in the body and various metabolic disorders caused by increased GH and insulin-like growth factor-1 (IGF1). Surgical treatment of pituitary tumors is the preferred standard of care, but only 40-70% of patients can be treated with surgical treatment alone. In many cases, complete resection of the tumor is not possible and the hormone imbalance persists after surgery. After surgical treatment, several additional treatments are needed to prevent hypersecretion of GH and to normalize blood levels of IGF-1.

As first-line treatment after surgical resection, there are typically drug therapy and radiation therapy. The most common used drugs are octreotide and lanreotide, which are growth hormone analogues. However, according to the recent guideline, the endocrine remission rate obtained from post-operative drug therapy is only 17-35%. Although clinical trials are underway for new drugs, the burden of expensive drug costs, recurrence during drug withdrawal, and drug side effects remains major drawbacks. There is a need for therapeutic intervention to reduce the dose and duration of therapy, to prevent tumor recurrence, and to achieve rapid endocrinologic remission.

Stereotactic radiosurgery (SRS), such as gamma knife radiosurgery, has been actively introduced worldwide to control residual pituitary tumors and has been applied to more than 200 cases of intractable acromegaly. The effect of SRS on endocrine remission in patients who did not receive endocrine therapy was confirmed in the literature. In a study of 136 patients who underwent preoperative radiotherapy followed by more than 5 years of follow-up, 65.4% of patients reported endocrine remission. According to the recently published meta-analysis, SRS showed 93-100% tumor growth control and size reduction within 5 to 10 years after surgery. The endocrinologic remission rate was reported to be 40-60% at 5 years.

To date, SRS has been recommended for the treatment of growth hormone - secreting pituitary tumors in cases where surgical removal is not feasible from the beginning or if drug treatment fails after surgical removal. Only the retrospective study of SRS was performed and no prospective study was conducted at all. However, many institutions already prefer preemptive SRS treatment for residual tumor after surgery and have been practiced in many patients. Therefore, prospective clinical trials are needed to establish the basis for upfront SRS and establish the treatment strategy for patients who do not have endocrine remission after surgical treatment of GH secretory pituitary tumor.

ELIGIBILITY:
Inclusion Criteria:

* Among patients with acromegaly due to growth hormone secreting pituitary adenoma who underwent primary surgical resection, patients who fail to achieve endocrinologic remission at 3 months after surgery.
* On brain MRI scan at 3months after surgery, residual tumor is confirmed by clinicians

  * the definition of endocrinologic remission

    1. random growth hormone level < 2.5 ug/L
    2. normalization of age-matched insulin growth factor-1 level

Exclusion Criteria:

* patients with contraindication of stereotactic radiosurgery; e.g. pregnancy or planning pregnancy, or claustrophobia
* recurrent pituitary adenoma
* limited life expectancy due to systemic disease; e.g. malignant tumor, genetic disease, and terminal stage of renal or hepatic failure
* disability to clinic visit due to postoperative complications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
endocrinologic remission | at 2 year after initial enrollment
  Achieving random growth hormone level below 2.5 ug/L and normalization of insulin-growth factor-1 level

SECONDARY OUTCOMES:
tumor size | 1 year interval
  maximum diameter of tumor
drug requirement dosage | at 3 months after initial enrollment and 6 months thereafter for 2 years
  daily total dose requirement (multiplied dose per injection by number of injections)
side effect | at 3 months after initial enrollment and 6 months thereafter for 2 years
  radiation induced and drug related side effects
performance status | at 3 months after initial enrollment and 6 months thereafter for 2 years
  modified Rankin scale; lower values represent a better outcome as followings: 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.

CONTACTS AND LOCATIONS:
Overall Officials: Doo0Sik Kong, MD,Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gheorghiu ML. Updates in outcomes of stereotactic radiation therapy in acromegaly. Pituitary. 2017 Feb;20(1):154-168. doi: 10.1007/s11102-016-0783-5. PMID 28210908
- [Background] Lee CC, Vance ML, Xu Z, Yen CP, Schlesinger D, Dodson B, Sheehan J. Stereotactic radiosurgery for acromegaly. J Clin Endocrinol Metab. 2014 Apr;99(4):1273-81. doi: 10.1210/jc.2013-3743. Epub 2014 Jan 28. PMID 24471574
- [Background] Shin SS, Tormenti MJ, Paluzzi A, Rothfus WE, Chang YF, Zainah H, Fernandez-Miranda JC, Snyderman CH, Challinor SM, Gardner PA. Endoscopic endonasal approach for growth hormone secreting pituitary adenomas: outcomes in 53 patients using 2010 consensus criteria for remission. Pituitary. 2013 Dec;16(4):435-44. doi: 10.1007/s11102-012-0440-6. PMID 23179961
- [Background] Giustina A, Chanson P, Kleinberg D, Bronstein MD, Clemmons DR, Klibanski A, van der Lely AJ, Strasburger CJ, Lamberts SW, Ho KK, Casanueva FF, Melmed S; Acromegaly Consensus Group. Expert consensus document: A consensus on the medical treatment of acromegaly. Nat Rev Endocrinol. 2014 Apr;10(4):243-8. doi: 10.1038/nrendo.2014.21. Epub 2014 Feb 25. PMID 24566817
- [Background] Hazer DB, Isik S, Berker D, Guler S, Gurlek A, Yucel T, Berker M. Treatment of acromegaly by endoscopic transsphenoidal surgery: surgical experience in 214 cases and cure rates according to current consensus criteria. J Neurosurg. 2013 Dec;119(6):1467-77. doi: 10.3171/2013.8.JNS13224. Epub 2013 Sep 27. PMID 24074496
- [Background] Katznelson L, Laws ER Jr, Melmed S, Molitch ME, Murad MH, Utz A, Wass JA; Endocrine Society. Acromegaly: an endocrine society clinical practice guideline. J Clin Endocrinol Metab. 2014 Nov;99(11):3933-51. doi: 10.1210/jc.2014-2700. Epub 2014 Oct 30. PMID 25356808